CLINICAL TRIAL: NCT04200326
Title: Real-life First Dose Effect of Fasenra in Patients With Severe Uncontrolled Asthma
Acronym: TWINKLE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D3250R00061
Record Dates: First submitted 2019-11-05; First posted 2019-12-16 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Severe Uncontrolled Asthma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This pilot study will use novel technologies to collect information about the patient experience before and early after starting Fasenra (benralizumab) as standard of care for severe uncontrolled asthma in a real-world setting, to determine how the experience changes over time. Any detection of an early, subjective first-dose effect in this pilot study will be further validated in a larger follow-up study.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE: Explore the use of novel technologies to detect early changes in quality of life (QoL) within the first 4 weeks after first dose of Fasenra for the treatment of severe uncontrolled asthma.

ENDPOINTS: Improvement in QoL measures, and physical and mental well-being as assessed by an increase in positive facial expressions, positive keywords, and quality of life biomarkers, with a decrease in asthma symptoms and improvement in FEV1 and PEF within the first 4 weeks after beginning Fasenra.

TARGET POPULATION: Individuals aged 18-75 years with severe asthma uncontrolled (ACQ >=1.5) on current medications (HD-ICS/LABA with/without other maintenance therapies except biologics). Patients beginning Fasenra asstandard of care as specified by NICE guidelines.

STUDY DURATION: The study duration per patient will be approximately 6 weeks from the enrolment visit to end of recorded data. Subjects will record data for 2 weeks prior to their first injection with Fasenra and then for 4 more weeks post-injection. PROCEDURESPatients will be required to visit the study site 3 times (enrolment and onboarding visit, Fasenra injection visit, last visit), and perform daily tasks at home in between site visits

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18-75 years with severe asthma uncontrolled (ACQ >=1.5) on current medications (HD-ICS/LABA with/without other maintenance therapies except biologics).
* Patients beginning Fasenra as standard of care as specified by NICE guidelines. That is, patients having either 4 exacerbations in the previous year and an eosinophil count over 300 cells/ microliter OR 3 exacerbations in the previous year and an eosinophil count over 400 cells/ microliter.
* Provision of informed consent prior to any study specific procedures
* Patients must have a smartphone that is compatible with the device software (iOS and Android).
* Availability of, and willingness to use, without reimbursement of any potential additional costs incurred, their computer and/or iOS/Android device for the collection and transmission of information
* English speaking and reading (ability to understand ICF, patient materials, the study app and to interact with the onboarding agent).

Exclusion Criteria:

* Patients taking daily prednisolone (or equivalent)
* Patients currently taking a biologic medication or participating in a clinical study involving a biologic medication for a respiratory illness.
* Comorbid conditions that cause symptoms similar to those experienced with asthma (e.g./ cough, wheeze, breathlessness, or nighttime awakening).
* Patients with comorbidities that also significantly affect patient's quality of life and daily functioning as determined by the treating physician.
* Presence of other chronic pulmonary conditions (e.g./ COPD)
* Patients that in the opinion of the physician are unlikely to complete 6 weeks of the study (example reasons: digital literacy, unwillingness/inability to interact with apps; historically poor adherence to study procedures)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals aged 18-75 years with severe asthma uncontrolled (ACQ >=1.5) on current medications (HD-ICS/LABA with/without other maintenance therapies except biologics) who are beginning Fasenra treatment as standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2020-04-09 (Actual); Study Completion 2020-04-09 (Actual)

PRIMARY OUTCOMES:
Sentiment score | 6 weeks from baseline
  Evaluate if the PROACT system can detect early signs of changes in quality of life (QoL) using sentiment analysis to determine changes in peoples' emotions as a subjective measure of first-dose effects of a medication. the score should be the positivity of the expression, scaled from 0 (the most negative) to 1.0 (totally positive).
Emotion confidence score | 6 weeks from baseline
  Evaluate if the PROACT system can detect early signs of changes in quality of life (QoL) using emotion confidence score to determine changes in peoples' emotions as a subjective measure of first-dose effects of a medication. Emotion confidence score should be the confidence (probability) of the predicted emotion given by the machine learning model. The scores will be scaled proportionally to have a sum of 1.0 for each frame of the video.
Key phrase extraction | 6 weeks from baseline
  Evaluate if the PROACT system can detect early signs of changes in quality of life (QoL) using key phrase extraction to determine changes in peoples' emotions as a subjective measure of first-dose effects of a medication. Key phrase extraction is a descriptive summary of the video message recorded.
Message analysis | 6 weeks from baseline
  Evaluate if the PROACT system can detect early signs of changes in quality of life (QoL) using message analysis to determine changes in peoples' emotions as a subjective measure of first-dose effects of a medication. The message analysis will define:
  The topic - what it is that the participant is trying to share. This is coded using an evolving, hierarchical, lexicon.
  The impact - if reported, the impact that this is having on the participant is also coded. An interpreted impact color scale (green-amber-red) is also applied by the analysts to aid quick identification of the most, and least, impactful things.
  The outcome - if reported, what the person did as a result of what happened. This is also coded so that it can also be aggregated across patients.

SECONDARY OUTCOMES:
PEF | 6 weeks
  Association between any onset of effect seen for PROACT measures and lung function (PEF, Peak Expiratory Flow) measurements. it can either be measured in L/sec or L/min .
FEV1 | 6 weeks
  Association between any onset of effect seen for PROACT measures and lung function (FEV1, Forced Expiratory Volume in 1 Second) measurements. Measured in liters.
FEV1/FVC | 6 weeks
  Association between any onset of effect seen for PROACT measures and lung function (FEV1/FVC (forced vital capacity), ratio of FEV1 to FVC ) measurements. Can be expressed as a percentage or ratio.
ACQ-6 Score | 6 weeks
  Association between any onset of effect seen for PROACT measures and PRO ACQ-6, using the ACQ-6 score. Patients are asked to recall how their asthma has been during the previous week by responding to 6 questions. Questions are weighted equally and scored from 0 (totally controlled) to 6 (severely uncontrolled). The mean ACQ-6 score is the mean of the responses. Mean scores of ≤0.75 indicate well-controlled asthma, scores between 0.75 and <1.5 indicate partly controlled asthma, and a score ≥1.5 indicates not well-controlled asthma.
SGRQ Score | 4 weeks from Fasenra injection
  Association between any onset of effect seen for PROACT measures and PRO SQRQ, using the SGRQ Score. The SGRQ is a 50-item PRO instrument developed to measure the health status of patients with airway obstruction diseases. The questionnaire is divided into 2 parts: part 1 consists of 8 items pertaining to the severity of respiratory symptoms in the preceding 4 weeks; part 2 consists of 42 items related to the daily activity and psychosocial impacts of the individual's respiratory condition.
  The SGRQ yields a total score and 3 domain scores (symptoms, activity, and impacts). The total score indicates the impact of disease on overall health status. This total score is expressed as a percentage of overall impairment, in which 100 represents the worst possible health status and 0 indicates the best possible health status. Likewise, the domain scores range from 0 to 100, with higher scores indicative of greater impairment.
daily UMotif measure | 6 weeks
  Association between any onset of effect seen in the daily uMotif measures and the ACQ-6 and SQRQ/lung function measurements will be assessed. The UMotif Quality of Life questionnaire consists of 10 separate 5 point Likert scale questions. Of these, 8 are required questions, and the remaining 2 are chosen at enrolment by patients from a choice of 4 possible questions. Responses to each of these questions will be compared to their own baseline at enrolment to derive personalized metrics. A composite metric will also be created by appropriately combining the individual question responses.
  The required 8 questions will be summarized descriptively by day. The 2 optional questions that patients report daily will be reported descriptively.

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Hagger, Study Director — Astra Zeneca R&D

REFERENCES:
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3250R00061&attachmentIdentifier=dd181143-1876-4f41-bda6-e7745459852e&fileName=D3250R00061_TWINKLE_Study_Report_Synopsis_11Mar2021_Redacted_V2.pdf&versionIdentifier=